CLINICAL TRIAL: NCT06869122
Title: Assessment of the Safety and Performance of the AB1 Electrosurgical System for Bronchoscopic Microwave Ablation of Lung Tissue in Surgical Candidates - UK
Brief Title: Bronchoscopic Microwave Ablation of Lung Tissue in Surgical Candidates - UK
Acronym: AB1MALTISC-UK
Status: Recruiting | Type: Observational
Sponsor: Creo Medical Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: PD-GTD-AB1UK-003
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Ablation; Microwave; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Resected lung tissue and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microwave ablation: Patients with a malignant lung nodule who are candidates for surgical resection.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Bronchoscopy and microwave ablation of the lung tumour prior to surgical resection.

SUMMARY:
This study involves the use of a medical device, the Creo Medical MicroBlate Flex instrument, to heat and destroy lung tumour cells using microwave energy (this is also called ablation). In this study, we are investigating whether the ablation instrument can be used effectively to treat lung tumours or tumours that have spread to the lungs. If successful, using this technology may mean future patients may not need to undergo surgical removal of these types of lung tumours.

The aim of this study is to evaluate the safety and performance of the MicroBlate Flex instrument in treating individuals with cancerous lung tumours that are due to be removed by surgery. All participants in the study will undergo the microwave ablation procedure, which is a separate and additional procedure to their surgical procedure.

The study, funded by Creo Medical, will be conducted at a single site in the UK, and will involve up to 18 participants.

DETAILED DESCRIPTION:
Participation (approximately 2 months) in this study, will include a screening visit, a bronchoscopy procedure that includes the microwave ablation treatment, and the planned surgical removal of the lung tumour 7 to 21 days after the ablation.

There are 2 follow-up visits, one at 7 days after the ablation treatment, the second just before the planned surgical procedure. After surgery, patients will be monitored according to the hospital's routine clinical practice. Participation in the research study ends once the patient is discharged from hospital.

Participation in this study has the potential to provide the following benefits for other people who have the same medical condition:

* The option of choosing microwave ablation as an alternative treatment for lung tumours and avoiding a major surgical procedure.
* Shorter patient recovery times.
* Reduced incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

Patients who:

1. Have signed informed consent.
2. Subject is willing and able to comply with all aspects of the treatment and evaluation schedule.
3. Are ≥ 18 years old.
4. Have lung lesion(s)/nodule(s) which are histopathological confirmed as cancer.
5. Have soft tissue lung lesion(s):

   * ≤ 20 mm in the largest dimension of the pulmonary window
6. Are candidates for surgical resection as determined by a multi-disciplinary team (MDT) or tumour board.
7. > 10 mm of tumour-free lung parenchyma between target tumour and pleura or fissure.
8. Subject is willing and able to comply with the study protocol requirements.
9. Are assigned an ASA (American Society of Anaesthesiologists) score of ≤ 3 or the patient is deemed fit for general anaesthesia.

Exclusion Criteria:

Patients who:

1. Have target nodule(s) within the International Association for the Study of Lung Cancer (IASLC) "Central Zone" (including bronchial tree, major vessels, heart, oesophagus, spinal cord, and phrenic & laryngeal nerves).
2. Are pregnant or breast feeding, as determined by standard site practices.
3. Have participated in an investigational drug or device research study within 30 days of enrolment that would interfere with this study.
4. Have a physical or psychological condition that would impair study participation or jeopardise the safety or welfare of the subject.
5. Have an expected survival less than 12 months.
6. Have an implantable device, including pacemakers or other electronic implants.
7. Have known pulmonary hypertension (PASP [pulmonary artery systolic pressure] >50mmHg).
8. Subject had a prior pneumonectomy.
9. Diagnosis of Small Cell Lung Cancer.
10. Subject had a therapeutic intervention (e.g., SBRT) within same lobe as the target lesion.
11. Subjects currently undergoing or underwent chemotherapy, systemic immunosuppressive treatment, or radiotherapy within 3 months of planned Study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population going through lung cancer screening at investigative site.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety of the MicroBlate Flex AB1 system in lung tumour ablation | Up to 21 days after the ablation procedure
  Identification of serious device-related adverse events associated with the delivery of microwave energy by the AB1 system from ablation (Day 0) up to the first surgical incision for the resection (Day 7-21)
Technical Success and Performance of the AB1 instrument | Up to 28 days post ablation procedure
  Initial technical success, defined as successful bronchoscopic access by the AB1 instrument of the target tissue, delivery of the scheduled microwave energy to the target tissue (per pre-specified target) and confirmed ablation as evidenced by macroscopic assessment post-surgical resection of the ablated lesion

SECONDARY OUTCOMES:
Assessment/visualization/quantification of the dimensions of the ablated tissue including assessment of margin relative to lesion | Up to 1 week post surgical resection procedure
  Dimensions of the ablated tissue to confirm, correct or add to the IFU-reported relationship between AB1 ablation time and dimensions and volume of the ablated tissue, per pre-specified target
Assessment/visualization/quantification of the dimensions of the ablation observed within the post-ablation CT | Up to 1 week post ablation procedure
  Dimensions of the ablated tissue as evidenced on the post-ablation CT
Procedural Time | Up to 1 week post ablation procedure
  Procedural time to be captured in the electronic case report form
Assessment of ease of system use (Clinician Questionnaires) | Up to 1 week post ablation procedure
  Questionnaires to be completed by clinicians following each procedure, rating their responses on a Likert scale of 1 to 7, with 1 being "extremely clear/easy" and 7 being "extremely difficult"

OTHER OUTCOMES:
Assessment of immunological response following microwave ablation procedure | Up to 28 days post ablation procedure
  Immunological response, as determined by change from baseline to pre-surgical resection in immunological and inflammatory blood markers

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Royal Brompton Hospital, Sydney Street, London, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Summary aggregate information will be published in a PRJA at the conclusion of the study.

REFERENCES:
- [Background] Chang et al The Lancet Oncology 2015 Vol 16, Issue 6, 630 - 637
- [Background] SABR UK Consortium. "Stereotactic Ablative Body Radiation Therapy (SABR): A Resource." Version 6.1. January 2019.
- [Background] Chen H, Senan S, Nossent EJ, Boldt RG, Warner A, Palma DA, Louie AV. Treatment-Related Toxicity in Patients With Early-Stage Non-Small Cell Lung Cancer and Coexisting Interstitial Lung Disease: A Systematic Review. Int J Radiat Oncol Biol Phys. 2017 Jul 1;98(3):622-631. doi: 10.1016/j.ijrobp.2017.03.010. Epub 2017 Mar 15. PMID 28581404
- [Background] Boffa DJ, Allen MS, Grab JD, Gaissert HA, Harpole DH, Wright CD. Data from The Society of Thoracic Surgeons General Thoracic Surgery database: the surgical management of primary lung tumors. J Thorac Cardiovasc Surg. 2008 Feb;135(2):247-54. doi: 10.1016/j.jtcvs.2007.07.060. Epub 2007 Dec 21. PMID 18242243
- [Background] Licker MJ, Widikker I, Robert J, Frey JG, Spiliopoulos A, Ellenberger C, Schweizer A, Tschopp JM. Operative mortality and respiratory complications after lung resection for cancer: impact of chronic obstructive pulmonary disease and time trends. Ann Thorac Surg. 2006 May;81(5):1830-7. doi: 10.1016/j.athoracsur.2005.11.048. PMID 16631680
- [Background] Covey AM, Gandhi R, Brody LA, Getrajdman G, Thaler HT, Brown KT. Factors associated with pneumothorax and pneumothorax requiring treatment after percutaneous lung biopsy in 443 consecutive patients. J Vasc Interv Radiol. 2004 May;15(5):479-83. doi: 10.1097/01.rvi.0000124951.24134.50. PMID 15126658